CLINICAL TRIAL: NCT02483351
Title: Aneurysmal Subarachnoid Hemorrhage: Red Blood Cell Transfusion and Outcome - A Pilot Randomized Controlled Trial
Brief Title: Aneurysmal Subarachnoid Hemorrhage: Red Blood Cell Transfusion and Outcome
Acronym: SAHaRA Pilot
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Shane English, Associate Scientist, Ottawa Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20150433-01H
Record Dates: First submitted 2015-06-25; First posted 2015-06-26 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2018-04

CONDITIONS: Subarachnoid Hemorrhage
Keywords: Blood Transfusion
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liberal RBC Transfusion Strategy (Experimental)
  Interventions: Other: Liberal Red Blood Cell Transfusion Strategy
- Restrictive RBC Transfusion Strategy (Active Comparator)
  Interventions: Other: Restrictive Red Blood Cell Transfusion Strategy

INTERVENTIONS:
Other: Liberal Red Blood Cell Transfusion Strategy — RBC Transfusion strategy with hemoglobin trigger of 100g/L
  Arms: Liberal RBC Transfusion Strategy
Other: Restrictive Red Blood Cell Transfusion Strategy — Optional RBC Transfusion with hemoglobin trigger of <=80g/L
  Arms: Restrictive RBC Transfusion Strategy

SUMMARY:
The purpose of this study is to determine the feasibility of conducting a large trial examining the effect on clinical outcome of a liberal red blood cell (RBC) transfusion strategy compared to a restrictive strategy (usual care) in patients with aneurysmal subarachnoid hemorrhage (SAH).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old at time of presentation
2. First ever episode aneurysmal SAH
3. Confirmed aneurysmal SAH diagnosis: as confirmed by treating Neurosurgeon or Neuro-interventionalist and supported by blood in subarachnoid space (demonstrated on cranial imaging or cerebrospinal fluid positive for xanthochromia) that is the result of a ruptured saccular aneurysm (confirmed by cranial imaging - cranial topography or magnetic resonance imaging angiography or catheter angiogram)
4. Incident hemoglobin ≤100g/L within 14 days following SAH (defined by first day of hospital presentation)

Exclusion Criteria:

1. Physician and or family decision to withdraw/withhold critical care at time of enrolment
2. Active bleeding with hemodynamic instability at time of enrolment
3. Patients with contra-indication or known objection to blood transfusions
4. SAH due to causes other than saccular aneurysm rupture including mycotic, traumatic and dissecting aneurysms, and aneurysms associated with arteriovenous malformations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-10; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Randomization Rate | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Shane English, MD MSc FRCPC, Principal Investigator — Ottawa Hospital Research Institute; Lauralyn McIntyre, MD MSc FRCPC, Principal Investigator — Ottawa Hospital Research Institute
Locations (3):
- Canada (3):
  - Vancouver General Hospital, Vancouver, British Columbia
  - Hamilton Health Sciences Centre, Hamilton, Ontario
  - Shane English, Ottawa, Ontario

REFERENCES:
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Fergusson DA, Pagano MB, Roubinian NH, Turgeon AF, Valentine S, Trivella M, Doree C, Hebert PC. Transfusion thresholds and other strategies for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2025 Oct 20;10(10):CD002042. doi: 10.1002/14651858.CD002042.pub6. PMID 41114449
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Trivella M, Roubinian N, Fergusson DA, Triulzi D, Doree C, Hebert PC. Transfusion thresholds for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2021 Dec 21;12(12):CD002042. doi: 10.1002/14651858.CD002042.pub5. PMID 34932836
- [Derived] English SW, Fergusson D, Chasse M, Turgeon AF, Lauzier F, Griesdale D, Algird A, Kramer A, Tinmouth A, Lum C, Sinclair J, Marshall S, Dowlatshahi D, Boutin A, Pagliarello G, McIntyre LA; Canadian Critical Care Trials Group. Aneurysmal SubArachnoid Hemorrhage-Red Blood Cell Transfusion And Outcome (SAHaRA): a pilot randomised controlled trial protocol. BMJ Open. 2016 Dec 7;6(12):e012623. doi: 10.1136/bmjopen-2016-012623. PMID 27927658